CLINICAL TRIAL: NCT03452189
Title: The Effect of an Antibiotic on the Production of Uremic Toxins by the Gut Microbiome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17-00963
Record Dates: First submitted 2018-01-23; First posted 2018-03-02 (Actual); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: randomized double-blinded placebo-controlled crossover study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 250mg of oral vancomycin First (Active Comparator): After 3 months, initial experimental group will be switched to placebo for 3 months.
  Interventions: Drug: Vancomycin; Other: Placebo
- Placebo First (Placebo Comparator): After three months, the control group will be crossed over to weekly oral vancomycin (250mg)
  Interventions: Drug: Vancomycin; Other: Placebo

INTERVENTIONS:
Drug: Vancomycin — Oral vancomycin 250mg capsules
  Other Names: vancomycin hydrochloride capsules
Other: Placebo — Placebo Pills distributed by Research Pharmacy labeled "placebo."

SUMMARY:
The purpose of this study is to determine if multiple doses of vancomycin over the course of 3 months will perturb the intestinal flora (microbiome) and result in reduced serum concentration of the uremic toxin indoxyl sulfate and p-cresyl sulfate. The design of the study will permit investigators to assess the variability of serum uremic retention solute concentrations with and without antibiotic over a three-month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable chronic kidney disease on hemodialysis with a fistula or an AV graft.

Exclusion Criteria:

* Antibiotics received within the last 3 months;
* recent diarrhea
* known allergy to vancomycin
* history of C. difficile infection
* elevation of white blood cell count or fever within one week of enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-08-18 (Actual); Study Completion 2018-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Lowenstein, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.

RESULTS

PARTICIPANT FLOW:
Groups:
- 250mg of Oral Vancomycin First, Then Placebo: 250mg of Oral Vancomycin given for 3 months then crossed over to placebo for additional 3 months (no washout period).
- Placebo First, Then 250mg of Oral Vancomycin: Placebo given for 3 months then crossed over to 250 mg of Oral Vancomycin for additional 3 months (no washout period).
Period: First Intervention (3 Months)
Arm/Group | 250mg of Oral Vancomycin First, Then Placebo | Placebo First, Then 250mg of Oral Vancomycin
Started | 10 | 5
Completed | 5 | 5
Not Completed | 5 | 0
Not completed — Adverse Event | 1 | 0
Not completed — insufficient samples of plasma and stool | 4 | 0
Period: Intervention 2 (3 Months)
Arm/Group | 250mg of Oral Vancomycin First, Then Placebo | Placebo First, Then 250mg of Oral Vancomycin
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo First or 250mg of Oral Vancomycin First (Crossover After 3 Months): Total cohort
Arm/Group | Placebo First or 250mg of Oral Vancomycin First (Crossover After 3 Months)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2
  Black | 3
  Asian | 2
  Hispanic | 6
  Other or more than one | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Concentration Measure of Indoxyl Sulphate (IS)
Description: Plasma concentrations of IS were measured by HPLC (high pressure liquid chromatography).
  Assessed weekly between day 0 and Week 4; change from baseline/day 0 to Week 4 reported
Time Frame: 4 weeks
Population: As there was no "washout period" following vancomycin, for the analysis of vancomycin effect, investigators compared the changes in solute levels in all 10 subjects while receiving vancomycin to the changes seen in the 5 "Z" series subjects while receiving placebo as the initial treatment.
Measure: Mean (Standard Deviation); unit: µM/ml
Arm/Group | 250mg of Oral Vancomycin First, Then Placebo | Placebo First, Then 250mg of Oral Vancomycin
Number analyzed (Participants) | 10 | 5
µM/ml | -25.31 (36.3) | 9.71 (49.80)

2. Primary Outcome: Change in Plasma Concentration Measure P-Cresyl Sulphate (PCS)
Description: Plasma concentrations of P-Cresyl Sulphate (PCS) were measured by HPLC (high pressure liquid chromatography)
  Assessed weekly between day 0 and Week 4; change from baseline/day 0 to Week 4 reported
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µM/ml
Arm/Group | 250mg of Oral Vancomycin First, Then Placebo | Placebo First, Then 250mg of Oral Vancomycin
Number analyzed (Participants) | 10 | 5
µM/ml | -73.51 (127.00) | 0.64 (79.50)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 250mg of Oral Vancomycin First | Placebo First
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT03452189/Prot_SAP_000.pdf